CLINICAL TRIAL: NCT03390140
Title: ReInventing Yourself After SCI: A Multi-site Randomized Controlled Trial of an Intervention to Improve Outcomes After Spinal Cord Injury
Brief Title: ReInventing Yourself After SCI: an Intervention to Improve Outcomes After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Craig Hospital (Other)
Collaborators: University of Michigan (Other); Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90DPHF0002-01-00
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; Group Intervention; Self Efficacy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (Experimental): ReInventing Yourself after SCI structured group CBT and ReInventing Yourself after SCI study-specific workbook
  Interventions: Behavioral: ReInventing Yourself after SCI structured group CBT; Behavioral: ReInventing Yourself after SCI study-specific workbook
- Indiv (Active Comparator): ReInventing Yourself after SCI study-specific workbook and ReInventing Yourself after SCI YouTube videos
  Interventions: Behavioral: ReInventing Yourself after SCI study-specific workbook; Behavioral: ReInventing Yourself after SCI YouTube videos
- Control (No Intervention): No group sessions, no YouTube videos, no workbook

INTERVENTIONS:
Behavioral: ReInventing Yourself after SCI structured group CBT — ReInventing Yourself after SCI intervention integrates positive psychotherapy concepts into structured group cognitive behavioral therapy (CBT) to develop optimistic self-efficacy beliefs, thereby strengthening resilience to emotional distress, enhancing a sense of well-being and promoting a more active lifestyle. The intervention consists of six weekly two-hour facilitator-led sessions that include didactic presentations of eight core skills and related experiential exercises with extensive group discussion.
  Arms: Group
Behavioral: ReInventing Yourself after SCI study-specific workbook — A study-specific workbook that incorporates positive psychotherapy concepts to develop optimistic self-efficacy beliefs, thereby strengthening resilience to emotional distress, enhancing a sense of well-being and promoting a more active lifestyle.
  Arms: Group; Indiv
Behavioral: ReInventing Yourself after SCI YouTube videos — YouTube videos containing the content of the ReInventing Yourself after SCI structured group CBT sessions
  Arms: Indiv

SUMMARY:
The primary goal of this study is to conduct a multi-site RCT to evaluate the replicability and efficacy of the ReInventing Yourself after SCI intervention in improving health and function outcomes for persons with spinal cord injury (SCI). A total of 252 participants will be randomized to one of three research arms: 1) Group treatment plus workbook (Group), 2) individual self-study through YouTube video plus workbook (Indiv), and 3) no treatment, no workbook (Control). Participants randomized to the Group arm will attend 6 virtual weekly group sessions led by a pair of group facilitators and will utilize the study workbook. Indiv arm participants will receive the workbook and will be instructed to independently access YouTube videos of the group session content. Control arm participants will not receive any intervention during the 6 week period. Participants in all three arms will be assessed at identical time points throughout the study: baseline, 6 weeks, 14 weeks, 22 weeks, 30 weeks, and 46 weeks.

It is hypothesized that individuals in the Group intervention arm will show greater improvements after the six week intervention in SCI-specific and general self-efficacy, emotional well-being, increased societal participation, less depressive and anxiety symptomatology, and improved resilience than participants in the Indiv and Control arms.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a multi-site randomized controlled trial (RCT) to evaluate the replicability and efficacy of a structured six-week, manualized, group therapy intervention, ReInventing Yourself after SCI that delivers positive psychology concepts within a cognitive behavioral therapy (CBT)-based model. The goals of this RCT are to increase SCI-specific and general self-efficacy, enhance emotional well-being, and improve participation in society for people with SCI living in the community. Craig Hospital is the lead site for this study, collaborating with the University of Michigan, Ann Arbor, and Kessler Institute for Rehabilitation in New Jersey.

The intervention is delivered through six sessions, each lasting approximately 2 hours. Eight skills are presented over the course of the intervention to address reframing a person's method of looking at events, building confidence by focusing on personal strengths, developing methods of recognizing and appreciating the good in one's life and expressing gratitude for positive attributes. These skills are presented in a specific sequence through a workbook so that participants can gain mastery of introductory concepts before undertaking those that are both more difficult and complex.

The RCT will have three research arms: 1) Group treatment plus workbook (Group), 2) individual self-study through YouTube video plus workbook (Indiv), and 3) no group or individual sessions, no workbook (Control). It is hypothesized that presenting the positive psychotherapy topics in an interactive structured CBT group format while restructuring maladaptive thought processes and providing experiential opportunities to reinforce behavioral change will result in increased self-efficacy, enhanced well-being and improved societal participation. Three specific hypotheses will be tested:

Hypothesis 1 (Primary): Individuals in the Group arm will show greater improvements after the six week intervention in SCI-specific and general self-efficacy, emotional well-being, increased societal participation, less depressive and anxiety symptomatology, and improved resilience than participants in the Indiv and Control arms.

Hypothesis 2 (Secondary): Individuals in the Group arm will maintain greater improvements through 46 weeks post-intervention in SCI-specific self-efficacy than participants in the Indiv and Control arms.

Hypothesis 3 (Secondary): Individuals in the Group arm will show greater improvements after six weeks of treatment and through 46 weeks post-intervention in general self-efficacy, life satisfaction, community participation, resilience, and less depressive and anxiety symptomatology than participants in the Indiv and Control groups.

The Moorong Self-Efficacy Scale (MSES) will serve as the primary outcome measure for this study. Secondary outcome measures include the General Self-Efficacy Scale, Diener Satisfaction with Life Scale, and measures of participation, resilience, anxiety and depression.

Each collaborating site will enroll 84 individuals to be randomized into one of the three study arms in waves of 21 people per wave (up to 6 waves per site). Training of site facilitators will take place at Craig Hospital.

ELIGIBILITY:
Inclusion Criteria:

* History of spinal cord injury/disorder (SCI/D) at any neurological level
* At least 4 weeks post-discharge from initial inpatient rehabilitation
* English speaking in order to complete study measures and participate in group interactions
* Access to the internet and a laptop/desktop computer/smartphone with webcam and the ability and willingness to download Zoom software to join a video conference
* Able to provide informed consent to participate.

Exclusion Criteria:

* Diagnosed with MS, Lupus, ALS, or Spina Bifida
* History of moderate or severe traumatic brain injury
* Current participation in another RCT
* Unable to verbally communicate
* Unable to attend group sessions
* Active participation in another formal clinical group or psychological therapy
* Currently experiencing moderately severe or greater levels of depressive symptoms which would require more intense treatment than is provided in this intervention, as evidenced by a score of 15 or higher on the PHQ-9
* Has any medical or psychological condition that, in the judgment of the investigators, precludes successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2018-07-22 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Moorong Self-Efficacy Scale (MSES) - assessing change over time | The MSES will be administered at baseline and subsequent follow-up assessments (i.e., 6 weeks, 14 weeks, 22 weeks, 30 weeks, 46 weeks)
  The MSES is a 16 item self-report measure of self-efficacy related to everyday life activities, designed specifically for persons with SCI. Individuals use a 7-point Likert scale ranging from 1 (very uncertain) to 7 (very certain) to rate their ability to perform 16 everyday tasks, with higher scores representing greater perceived self-efficacy. A Total Score, ranging from 16 to 112 is calculated by summing all item responses

SECONDARY OUTCOMES:
Generalized Self-Efficacy Scale (GSES)- assessing change over time | The GSES will be administered at baseline and subsequent follow-up assessments (i.e., 6 weeks, 14 weeks, 22 weeks, 30 weeks, 46 weeks)
  The GSES is a questionnaire designed to assess a person's ability to cope with a variety of difficult demands in life, with ten items scored using a Likert rating scale, ranging from 1 (not at all true) to 4 (exactly true).
Diener Satisfaction with Life Scale (SWLS)- assessing change over time | The SWLS will be administered at baseline and subsequent follow-up assessments (i.e., 6 weeks, 14 weeks, 22 weeks, 30 weeks, 46 weeks)
  The SWLS will be used to measure global life satisfaction. This is a five item measure on which respondents rate their life satisfaction using a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). A Total Score is calculated by summing each of the items, and has a range of 5 to 35, with higher scores representing greater perceived QoL.
Participation Assessment with Recombined Tools - Objective (PART-O)- assessing change over time | The PART-O will be administered at baseline and subsequent follow-up assessments (i.e., 6 weeks, 14 weeks, 22 weeks, 30 weeks, 46 weeks)
  The PART-O is a 24-item assessment of participation and has demonstrated good psychometric properties in measuring participation for people living with disabilities. An Averaged Total Score is computed by taking the mean of 17 items, with scores ranging from 0 (never participate in these types of activities) to 5 (almost always participate in these types of activities), with higher scores representing greater participation. This assessment will be utilized to measure overall participation.
Patient Health Questionnaire - 9 (PHQ-9)- assessing change over time | The PHQ-9 will be administered at baseline and subsequent follow-up assessments (i.e., 6 weeks, 14 weeks, 22 weeks, 30 weeks, 46 weeks)
  The PHQ-9 is a 9 item scale that will be used to assess depression. Respondents rate the frequency at which specific problems have been bothersome during the past two weeks, using a four point scale ranging from 0 (not at all) to 3 (nearly every day). A Total Score is calculated by summing all items, with higher scores indicating an increasing severity of depression.
General Anxiety Disorder 7-item (GAD-7)- assessing change over time | The GAD-7 will be administered at baseline and subsequent follow-up assessments (i.e., 6 weeks, 14 weeks, 22 weeks, 30 weeks, 46 weeks)
  The GAD-7 is a brief 7 item measure that will be used to assess the severity of general anxiety. Using a four point Likert scale ranging from 0 (not at all sure) to 3 (nearly every day), respondents rate how often they have been bothered by specific symptoms during the past two weeks. A Total Severity Score, ranging from 0 to 21, is calculated by summing all items.
The Connor-Davidson Resilience Scale (CD-RISC 10) short form- assessing change over time | The CD-RISC 10 will be administered at baseline and subsequent follow-up assessments (i.e., 6 weeks, 14 weeks, 22 weeks, 30 weeks, 46 weeks)
  The CD-RISC 10 will be used to measure resilience. The measure consists of 10 items using a 5-point Likert scale ranging from 0 (not true at all) to 4 (true nearly all of the time). The scale measures how the participant felt over the past month. The questionnaire produces an overall resilience score that ranges from 0-40, with higher scores representing greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Charlifue, PhD, Principal Investigator — Craig Hospital
Locations (3):
- United States (3):
  - Craig Hospital, Englewood, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - Kessler Foundation, West Orange, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided